CLINICAL TRIAL: NCT01392664
Title: TVTO Versus TVTFFM for Urinary Stress Incontinence
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, menahem neuman, Principal Investigator, Western Galilee Hospital-Nahariya
Other Study IDs: 920090040
Record Dates: First submitted 2011-06-29; First posted 2011-07-12 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Urinary Stress Incontinence Treated by TVT

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Women who had urinary stress incontinence and underwent one of two procedures: the classic TVTO or the Folke-Flam method of surgical operation, will be evaluated and compared.

DETAILED DESCRIPTION:
We will enroll women that underwent one of the two surgeries: TVTO or the modification where the needle passes somewhat to the side to prevent the post operative pain, for urinary stress incontinence. Data will be collected from the charts. Telephone interviews will be carried out. Physical examination will also be incorporated.

ELIGIBILITY:
Inclusion Criteria:

* Women with Urinary Stress Incontinence treated by TVT

Exclusion Criteria:

* Women without with Urinary Stress Incontinence or not treated by TVT

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with Urinary Stress Incontinence treated by TVT
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-02; Primary Completion 2013-02 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Resolution of urinary stress incontinence | One year after surgery
  We will question the women as for they have stress urinary incontinence. Physical examination data will also be retrieved.

SECONDARY OUTCOMES:
Side effect of surgery | six-12 months
  We will question the women if they have symptoms such as pain in the hip joints, vaginal discharge and bleeding. Physical examination will be retrieved from the charts.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Department of Obstetrics and Gynecology, Western Galilee Hospital, Nahariya
  - Clinics of Dr Neuman, Tel Aviv